CLINICAL TRIAL: NCT05983289
Title: A Single Center, Randomized, Double-blind, Placebo-controlled Study To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Single Escalating Doses Of HSK7653 In Healthy Subjects
Brief Title: Single Escalating Dose Study Of HSK7653 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HSK7653-101
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK7653 (Experimental): Single dose, oral
  Interventions: Drug: HSK7653
- Placebo (Placebo Comparator): Single dose, oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK7653 — HSK7653 tablets in six doses beginning at 5 mg and rising to 150 mg
  Arms: HSK7653
Drug: Placebo — Matching placebo tables in six doses beginning at 5 mg and rising to 150 mg
  Arms: Placebo

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) characteristics of single dose of HSK7653 tablets in healthy adult subjects, and to identify the metabolites of HSK7653 in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and Age ≤60 years
* BMI ≥18 and BMI ≤ 25 kg/m2 (Body Mass Index)
* Able to understand the procedures of the study, provide written informed consent, and be willing to comply with the protocol of the study

Exclusion Criteria:

* Any finding of the medical examination (physical examination, laboratory examination, 12-ECG, abdominal B-ultrasonography, etc) deviating from normal and of clinical relevance during screening
* Evidence or history of clinically significant renal, gastrointestinal (including pancreatitis), hepatic disease at the time of screening
* Has a positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), Treponema pallidum antibody (TP-Ab) or human immunodeficiency virus (HIV)
* Treatment with an investigational drug within 3 months
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception for the duration of the study and for at least 6 months after the last dose

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | First dose of study drug up to 29 days after last dose of study drug
  Assessment by adverse event monitoring, 12 lead ECGs, vital signs and laboratory measurements.

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration | Pre dose and at 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 72, 168 (day 8), 336 (day 15), 504(day 22), 672 (day 29) hours following single dose administration;
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Maximum Observed Plasma Concentration (Cmax) | Pre dose and at 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 72, 168 (day 8), 336 (day 15), 504(day 22), 672 (day 29) hours following single dose administration;
  Maximum Observed Plasma Concentration (Cmax)
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Pre dose and at 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 72, 168 (day 8), 336 (day 15), 504(day 22), 672 (day 29) hours following single dose administration;
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Plasma Decay Half-Life (t1/2) | Pre dose and at 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 72, 168 (day 8), 336 (day 15), 504(day 22), 672 (day 29) hours following single dose administration;
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Inhibition Rate of Dipeptidyl Peptidase 4 (DPP4) Activities following single dose administration | Pre dose and at 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 72, 168 (day 8), 336 (day 15), 504(day 22), 672 (day 29) hours following single dose administration;
  Inhibition Rate of Dipeptidyl Peptidase 4 (DPP4) Activities following single dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhong Liu, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No